CLINICAL TRIAL: NCT01589744
Title: Vacuum Device for Hemostasis in Obstetrics and Gynecology: Proof of Concept Study in the Post Partum Hemorrhage
Brief Title: Proof of Concept Study of a Sucker Hemostatic Intra Uterine in Postpartum Hemorrhage After Abruptio Placenta Assisted
Acronym: HEMOGYN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Non adequation between the medical device and the study population
Sponsor: AdministrateurCIC (Other)
Responsible Party: Sponsor-Investigator, AdministrateurCIC, principal investigator, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: DCIC 11 24
Record Dates: First submitted 2012-04-25; First posted 2012-05-02 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: No Placental Abruption; No Hemorrhage
Keywords: medical device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Suction cup Hemostatic Intra-Uterin (Experimental): The suction haemostatic cup will be positioned into the uterus, and the aim is to stop haemorrhage
  Interventions: Device: Suction cup Hemostatic Intra-Uterine, device not marked CE (not marketed)

INTERVENTIONS:
Device: Suction cup Hemostatic Intra-Uterine, device not marked CE (not marketed) — The haemostatic intra-uterine suction-cup is introduced in uterus and a depressure in this device is applied. This medical device is used for 5 minutes at maximum.

SUMMARY:
The postpartum hemorrhage (PPH) is the major complication of the delivery. In clinical practice, if after giving birth, the placenta is not expelled naturally, an active management should be triggered. Escalating therapy after obstetric maneuvers (placenta, uterus, examination of the birth canal), begins with uterotonic treatments for invasive treatments lead to embolization, vessel ligation and hysterectomy. However, the morbidity of these techniques and the desire to preserve fertility required to devise new therapeutic solutions, which have recently led to the development of an innovative medical device intrauterine hemostasis.

The postpartum haemorrhage are mainly the result of weak and bleeding from the surface corresponds to the placental insertion, which is no longer localized. With the innovative medical device, our main hypothesis is that the uterine walls will append to the walls of the cup after depressurization of the latter. The actuation of the suction cup will lead to aspiration of all sides of the uterus (it is mostly the anterior and posterior that are important). The suction cup is flexible to adapt to the size of the uterus in order to be placed and removed easily from the uterine cavity.

DETAILED DESCRIPTION:
In this study, as a first pass in Human, innovative medical device not CE marked, we did not aim to show control of the bleeding stops in the case of PPH but to prove, in a clinical situation with no foreseeable risk to the volunteers included (volunteers who have given birth without placental abruption after 30 minutes despite the directed delivery), proof of concept of using this system in these women that creates a vacuum in the Intra uterine Haemostatic vacuum and thus a joining of the walls of the uterus. This first step seems essential in order to effectively implement this medical device with serenity in emergency situations of PPH.

ELIGIBILITY:
Inclusion Criteria:

* woman between 18 and 45 years old,
* affiliation to the French social security system or equivalent,
* volunteers signed a consent to participate,
* volunteer is under loco-regional anaesthesia,
* volunteer whose the placenta has not taken off after 30 minutes despite the directed delivery.

Exclusion Criteria:

* volunteer carries uterine malformations,
* volunteer with post-partum haemorrhage (blood loss> 500 ml),
* volunteer allergic to silicon,
* volunteer under general anaesthesia,
* pregnancy not unique,
* volunteer with fever or suspected infection during labor,
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent
* Person under legal protection
* Person hospitalized for psychiatric care

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Number of participants for which there is a joining of the walls of the uterus around the suction cup after the depressurization. | 18 month
  Comparison of ultrasound images before and after depression in the suction cup. The joining of tissues on the suction cup is characterized by a better visualization of posterior structures following the depressurization by eliminating air in the haemostatic intra-uterine suction cup.

SECONDARY OUTCOMES:
Number of participants for which the setting up of the suction cup in uterus is a successful. | 18 month
  Qualification of success or failure of the setting up and score between 0 and 10 on a Visual,quantitative satisfaction scale.
Number of participant for which there is a persistence of the joining walls of the uterus around the suction cup between 1 and 5 minutes at maximum after passage of the depression with Redon Drainobag®. | 18 month
Number of participants for which the withdrawal of the suction cup from the uterus is a successful. | 18 month
  Qualification of success or failure of natural withdrawal of the suction cup and score between 0 and 10 on a visual, quantitative satisfaction scale.

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Equy, MD, Principal Investigator — Clinic of Gynecology and Obstetrics, University Hospital Grenoble - France
Locations (1):
- University Hospital Grenoble, Grenoble, France

REFERENCES:
- See also: Related Info — http://www.cic-it-grenoble.fr/